CLINICAL TRIAL: NCT02807896
Title: Multiple Biomarker Development Through Validation of Useful Markers Generated by Next Generation Bio-data Based Genome Research and Cohort Study
Brief Title: Validation of Useful Markers Generated by Next Generation Bio-data Based Genome Research and Cohort Study
Acronym: miRNA_Chip
Status: Completed | Type: Observational
Sponsor: CHANGHEE LEE (Industry)
Collaborators: Purdue University (Other); LG Electronics Inc. (Industry)
Responsible Party: Sponsor-Investigator, CHANGHEE LEE, Chief Research Engineer, LG Electronics Inc.
Organization: LG Electronics Inc. (Industry)
Other Study IDs: miRNA_Chip
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: BCL2 Gene mRNA Overexpression
Keywords: biomarker; pancreatic cancer; bile duct cancer; miRNA
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Among patients with pancreatic cancer or bile duct cancer without previous chemotherapy or radiation therapy, the subjects are divided into operable patients and inoperable patients.
  For operable patients, about 10cc (paxgene tube) of blood sample is collected before operation. After operation, 400mg of cancerous tissue and 400mg of normal tissue are requested and received from the gene bank of Severance Hospital where the tissues are stored.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- pancreatic cancer: pancreatic cancer 88
- bile duct cancer: bile duct cancer 101
- stomach cancer: stomach cancer 9
- colon cancer: colon cancer 5
- normal group: normal group 29

INTERVENTIONS:
Other:  — This study is cohort.

SUMMARY:
Multiple biomarker development through validation of useful markers generated by next generation bio-data based genome research and cohort study

DETAILED DESCRIPTION:
1. Objectives The study will be performed to develop the integrated analytical methods of genomic data and clinical data and the bio-control network analysis, through which knowledge-based integrated analysis system can be developed and then biomarker for early diagnosis and treatment of pancreatic cancer and bile duct cancer, and finally the customized disease management system. Also, it is to confirm the effectiveness of diagnostic chip for research purpose by applying pancreatic/bile duct cancer-specific biomarker, miRNA, found through the integrated analysis of genomic data and clinical data of patients with pancreatic/bile duct cancer to the blood of patients with pancreatic/bile duct cancer.
2. Effective evaluation method

The discrimination and calibration for algorithm through the diagnostic chip of each cancer type will all be examined using 10-fold cross-validation (100 repetitions). In the 10-fold cross-validation, the data is randomly divided into 10 same sized data, among which 9 are used in making a model for training and the remaining 1 is applied for test, and this process is randomly and independently repeated for 100 times.

The 10-fold cross-validated AUC is calculated to see the discrimination of diagnostic chip of each cancer type, and the 95% confidence interval is presented by non-parametric method.

The 10-fold cross-validated calibration plot is presented to see the calibration of diagnostic chip of each cancer type. The calibration plot visually demonstrate the degree of prediction by comparing the prediction probability of each group and the ratio of actual cancer patients after listing the prediction probability in the order and dividing it with regular intervals.

Then, for the same subjects, the AUC of the CA 19-9, the existing cancer diagnostic tool, is calculated and the 95% confidence interval is presented. To compare the diagnostic chip of each cancer type and the AUC of CA 19-9, p-value is calculated by non-parametric method of 10-fold cross-validated AUC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically diagnosed pancreatic cancer or bile duct cancer
* Patient age: 20~80 years old
* Patients who voluntarily determined to participate in the clinical trial and signed the informed consent for compliance
* Korean race

Exclusion Criteria:

* Patients with previous history of chemotherapy or radiation therapy for pancreatic cancer and/or bile duct cancer
* Patients who had treatment or surgery for cancer of other organ within 5 years before the clinical trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The number of target subjects and calculation basis for blood samples used in the development of multiple biomarker and diagnostic chip production are as below.
  Number of study subjects: 232 patients (pancreatic cancer 88, bile duct cancer 101, stomach cancer 9, colon cancer 5, normal group 29)
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2016-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
AUC(area under curve) | within 1week
  The AUC(area under curve) is calculated as an index for discrimination to see how well it discriminates algorithm through diagnostic chip for each cancer type.
  The calibration plot will be presented for the evaluation of calibration to see how well it calibrates algorithm through diagnostic chip for each cancer type, and the comparison of CA 19-9 by each cancer type and AUC differences of the diagnostic chip will be evaluated.

SECONDARY OUTCOMES:
cut-off of each biomarker, accuracy | within 1week
  The cut-off of each biomarker expression for maximizing the discrimination of diagnostic chips is calculated and presented as an index for analytical sensitivity.
  The accuracy considering the characteristics of diagnostic chip is calculated and presented.

CONTACTS AND LOCATIONS:
Overall Officials: Si Young Song, M.D. PhD, Principal Investigator — Severance Hospital, Yonsei University
Locations (1):
- Severance Hospital, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No